CLINICAL TRIAL: NCT06805656
Title: Multi Interventional Approaches to Mitigate HIV Reservoirs Aiming the Sustained HIV Remission Without Use of Antiretrovirals
Brief Title: Multi Interventional Approaches to Mitigate HIV Reservoirs Aiming the Sustained HIV Remission Without Antiretrovirals
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Ricardo Sobhie Diaz, Associated Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARC-11
Record Dates: First submitted 2022-03-25; First posted 2025-02-03 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hiv; HIV I Infection
Keywords: Dendritic Cell vaccination; antiretroviral intensification; Auranofin; Histone Deacetylase Inhibitor; residual viral replication; HIV sanctuaries; HIV latency
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; dolutegravir; lentiviral minigene vaccine of COVID-19 coronavirus; Auranofin; Niacinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antiretroviral Treated (ART) Group (No Intervention): Ten patients will receive no further intervention (control group)
- ART Intensification Group (Experimental): Sixty patients will be included in this stage to undergo the same interventions as Group 6 of the study under registration NCT02961829 of clinicaltrials.gov (antiretroviral intensification with dolutegravir and the Sirtuin Histone deacetylase inhibitor nicotinamide for 48 weeks, and gold salt for 24 weeks and dendritic cell vaccine.), with the adjustment to use also the maraviroc during the first 44 weeks.
  Interventions: Drug: Maraviroc; Drug: Dolutegravir; Biological: Dendritic Cell Vaccine; Drug: Auranofin; Drug: Sirtuin Histone deacetylase inhibitor

INTERVENTIONS:
Drug: Maraviroc — antiretroviral intensification
  Other Names: Selzentry; Celsentri
  Arms: ART Intensification Group
Drug: Dolutegravir — antiretroviral intensification
  Other Names: Tivicay
  Arms: ART Intensification Group
Biological: Dendritic Cell Vaccine — therapeutic vaccination
  Other Names: DC Vaccine
  Arms: ART Intensification Group
Drug: Auranofin — purging
  Other Names: Gold Salt
  Arms: ART Intensification Group
Drug: Sirtuin Histone deacetylase inhibitor — latency disruption
  Other Names: Nicotinamide
  Arms: ART Intensification Group

SUMMARY:
A modern and urgent challenge in fighting HIV infection is to achieve sustained HIV remission without the use of antiretrovirals. The investigators' preliminary data indicate that the use of combined strategies to mitigate the HIV proviral reservoir size among individuals with suppressive antiretroviral treatment achieved unprecedented results in the reduction of HIV DNA present in these cells and in the reduction of CD4 + and CD8 + T cell activation. Combined interventions include intensified antiretroviral treatment to mitigate residual HIV replication, use of a histone deacetylase inhibitor to interrupt viral latency, use of an anti-proliferative medication to reduce long-lived T cells that harbor HIV and a personalized dendritic cell therapy vaccine to eliminate cells with latent HIV infection or cells present in viral sanctuaries. Due to the good results obtained in the exploratory stage of the project, the investigators propose to expand it by recruiting a larger number of patient to confirm the previously obtained results and to generate new insights related to the mechanisms involved in viral latency, latency disruption and the effects of analytical treatment interruption of antiretrovirals among patients undergoing all above mentioned interventions.

ELIGIBILITY:
Inclusion Criteria:

- > 18 years old < 65 years old Documented HIV-1 infection. Has voluntarily signed ICF. On HAART ≥ 2 years, without changes in the 24 weeks immediately prior to screening.

HIV viral load <50 copies/mL, and never > 50 copies/mL on 2 consecutive occasions in the last 2 years. CD4 count nadir.

> 350 cells/ mm3 Current CD4 count > 500 cells/ mm3. R5 HIV-1 at Screening as defined by proviral DNA genotropism.

Exclusion Criteria:

- Any evidence of an active AIDS-defining condition. Any significant acute medical illness in the past 8 weeks. Women who are pregnant or breastfeeding. Use of any of the following within 90 days prior to entry: systemic cytotoxic chemotherapy; investigational agents; immunomodulators (colonystimulating factors, growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons); coumadin, warfarin, or other coumadin derivative anticoagulants. Use of an agent definitely or possibly associated with effects on QT intervals: amiodarone, arsenic trioxide, astemizole, bepridil, chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide, dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, probucol, procainamide, quinidine, sotalol, sparfloxacin, terfenadine, thioridazine.

Receipt of compounds with HDAC inhibitor-like activity, such as valproic acid or nicotinamide within the last 30 days. Potential participants may enroll after a 30-day washout period.

Known hypersensitivity to the components of gold salt, nicotinamide or its analogs.

Hepatitis B (HBsAg +) or Hepatitis C (HCV RNA +) infection. Known renal insufficiency defined as calculated creatinine clearance (Cockcroft Gault formula) <60 mL/min.

Subjects with a laboratory abnormality grade 3 or 4 with the following exceptions: pancreatic amylase, cholesterol, triglyceride, gamma glutamyl transpeptidase, bilirubin.

Any condition which, in the investigators opinion, could compromise the subject's safety or adherence to the trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Evolution of viral load of HIV RNA over the time frame of study | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Viral load count by qPCR at each time point to measure the viral persistence in each participant
Evolution of total DNA and episomal HIV in PBMCs | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Quantification of total DNA and episomal HIV in a virological assay
Evolution of cell-associated HIV RNA in PBMCs over the study time frame | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Quantification of HIV RNA in PBMCs by qPCR
Evolution of total DNA and episomal HIV DNA in lymphoid tissue (rectal biopsy) | baseline, week 48, after resurgence of viremia in the analytical interruption of antiretrovirals, or after 24 and 96 weeks after analytical interruption of antiretrovirals.
  Quantification by in-house virological assay
Evolution of the HIV DNA sequence of the V3 region of gp 120, protease, reverse transcriptase and integrase regions of the pol gene, and of the gag gene | baseline, week 24, week 48, after resurgence of viremia after ATI and before reintroduction of ART
  NGS sequencing of the V3 region of gp120, the protease, reverse transcriptase, and integrase regions of the pol gene, and of the gag gene of HIV DNA
Evolution of the HIV RNA sequence of the V3 region of gp 120, protease, reverse transcriptase and integrase regions of the pol gene, and of the gag gene | baseline, week 24, week 48, after resurgence of viremia after ATI and before reintroduction of ART
  NGS sequencing of the V3 region of gp120, the protease, reverse transcriptase, and integrase regions of the pol gene, and of the gag gene of HIV RNA
Evolution of CD4 + and CD8 + T lymphocyte count | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to a total of 36 months after ATI.
  Count by flow cytometry of CD4+ and CD8+ lymphocytes
Evolution of percentages of CD38 and HLA DR in CD4 + and CD8 + T lymphocytes | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Measurement by flow cytometry of cell activation of CD4+ and CD8+ T lymphocytes as a means of assessing immune and inflammatory responses
Evolution of plasma cytokines IL-2, IL-4, IL-6, IL-10, IL-17, TNF and IFN-γ | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Measurement by ELISA Assay of plasma cytokines IL-2, IL-4, IL-6, IL-10, IL-17, TNF and IFN-γ as a means of assessing immune and inflammatory responses
Changes in bacterial translocation levels by quantification of plasma LPS levels | baseline, weeks 12, 24, 36 and 48 and every 3 weeks after the antiretroviral ATI up to 36 months after antiretroviral ATI
  Assay for determining the proinflammatory level of endotoxin (LPS)

CONTACTS AND LOCATIONS:
Locations (1):
- CCDI, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
Because of the range of personal data gathered, IPD will be shared on request when properly anonymized.